CLINICAL TRIAL: NCT07280299
Title: A Randomized, Placebo-controlled, Double-blind, Phase 2a Study to Evaluate the Clinical Efficacy, Safety, Tolerability, and Biomarker Effects of 2 Dose Levels of GT-02287 in Participants With Early Parkinson's Disease
Brief Title: Efficacy, Safety, Tolerability, and Biomarker Effects of GT-02287 in Early Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gain Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GANX-001-V103
Record Dates: First submitted 2025-11-24; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — licorice extract - magnesium aluminometasilicate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose GT-02287 (Active Comparator): GT-02287 400 or 600 mg/day
  Interventions: Drug: Low Dose GT-02287
- High Dose GT-02287 (Active Comparator): GT-02287 800 or 1000 mg/day
  Interventions: Drug: High Dose GT-02287
- Placebo (Placebo Comparator): Magnesium aluminometasilicate (MAS)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Dose GT-02287 — Sachets containing 400 mg/day or 600 mg/day of active (GT-02287), depending on the participant's body weight. Each daily dose will be prepared as an oral suspension by mixing the content of 1 sachet with the vehicle (supplied in an amber glass bottle) and the requisite volume of tap water.
  Other Names: GT-02287 400 or 600 mg/day
  Arms: Low Dose GT-02287
Drug: High Dose GT-02287 — Sachets containing 800 mg/day or 1000 mg/day of active (GT-02287), depending on the participant's body weight. Each daily dose will be prepared as an oral suspension by mixing the content of 1 sachet with the vehicle (supplied in an amber glass bottle) and the requisite volume of tap water.
  Other Names: GT-02287 800 or 1000 mg/day
  Arms: High Dose GT-02287
Drug: Placebo — Sachets containing 420 to 1200 mg of MAS indistinguishable from the active sachets. Each daily dose will be prepared as an oral suspension by mixing the content of 1 sachet with the vehicle (supplied in an amber glass bottle) and the requisite volume of tap water.
  Other Names: Magnesium aluminometasilicate (MAS)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy, the safety, and the effect on biomarkers of 2 dose levels of oral GT-02287 over placebo after 48 weeks of treatment in treated and untreated participants with early PD.

DETAILED DESCRIPTION:
This is a 48-week, double-blind, randomized, placebo-controlled Phase 2a study testing two doses of oral GT-02287 in people with early Parkinson's disease (PD), both treated and untreated.

The study has three parts:

* Screening Period lasting up to 45 days
* Treatment Period lasting about 341 days
* Follow-up Period lasting up to 33 days Participants will have 7 onsite visits for efficacy, safety, tolerability, and biomarker assessments (Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, and a Follow-Up Visit at Week 52). In addition, there will be 5 additional visits for laboratory blood tests (Weeks 2, 16, 20, 30, and 42).

Approximately 111 participants will be randomized into three groups (high dose, low dose, placebo).

Participants can have idiopathic PD or be heterozygous for a pathogenic variant in the GBA1 gene. Participants who have other PD-associated genetic variants (e.g., leucine rich repeat kinase 2 [LRRK2]) are ineligible. All participants will be genotyped to determine their PD-associated genetic status before enrollment.

At the start, participants undergo screening and baseline tests, including motor assessments, quality of life, sensor measurements, and collection of fluid and blood samples for biomarkers. Some baseline tests may be done just before dosing.

The study will measure efficacy through various motor, quality of life, disease progression, non-motor and other symptoms of PD, and cognitive tests, along with wearable sensor data.

Safety will be assessed by recording adverse events, lab tests, vital signs, body weight, heart monitoring, and questionnaires.

The study will also analyze GT-02287 levels in blood and spinal fluid, and its effects on biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent and willing to comply with the requirements and restrictions of the study
* Willing to undergo PD-related genetic testing and analysis
* Any sex, ≥30 and ≤85 years of age
* Body mass index of ≥18 and ≤40 kg/m2 and a body weight of at ≥55 kg and <120 kg at Screening
* Diagnosis of PD based on MDS criteria
* Within 5 years of PD diagnosis
* Positive SAA in CSF at Baseline
* Hoehn & Yahr 1-2.5, inclusive
* Naïve to pharmacological treatment for PD with no initiation of dopaminergic treatment expected during the first 9 months of the study or on stable PD medication for ≥3 months prior to Screening, including ≥4 weeks at the same dose(s) immediately before Screening with no changes to dose(s), or medication(s) expected during the first 9 months of the study
* Not pregnant or breastfeeding
* If participant is either of childbearing potential or produces potentially viable sperm, participant must agree to use 2 forms of contraception (barrier method and a second highly effective form of birth control/contraception, as defined in the protocol) if engaging in potentially reproductive intercourse (with a partner who produces potentially viable sperm or is of childbearing potential, respectively)
* Agreeing not to participate in another investigational study while taking part in this study

Exclusion Criteria:

* Other neurological disorders, including but not limited to Alzheimer's disease, amyotrophic lateral sclerosis, frontotemporal dementia, progressive supranuclear palsy, corticobasal syndrome, Huntington's disease, multiple system atrophy, dementia with Lewy bodies, secondary (e.g. drug-induced) parkinsonism, multiple sclerosis, or epilepsy
* PD-associated LRRK2 pathogenic variant or other PD-associated genetic mutations other than GBA1
* Severe motor fluctuations and/or disabling dyskinesias based on the investigator's clinical assessment
* Deep-brain stimulation
* Hallucinations, delusions, or other psychotic symptoms requiring antipsychotic medication Use of dopamine antagonists (antipsychotics) or anticholinergic medications
* Dementia by clinical diagnosis and/or a MoCA score of ≤20 and/or a history of behavioral impairment
* Hypersensitivity to GT 02287 or any of its excipients
* Concomitant medications including drugs metabolized primarily by CYP3A4 that have a narrow therapeutic window, substrates of BCRP that have a narrow therapeutic window, strong or moderate inhibitors or strong inducers of CYP3A4 that could affect the metabolism and plasma levels of GT 02287, including herbal supplements and certain foods.
* Concomitant disease including, but not limited to cardiovascular conditions, diabetes, autoimmune disease, cancer, active infectious disease, psychotic disorders and symptoms, depressive symptoms, drug and/or alcohol misuse as defined in the protocol
* Clinically significant abnormalities in laboratory test
* Contraindications to lumbar puncture (LP) including current treatment with anticoagulants or any other contraindications that might preclude safe completion of the LP
* Blood donation >500 mL within 3 months
* Malabsorption or relevant disorder which may impact the absorption of GT-02287
* Participation in any interventional clinical study within 3 months or 5 half-lives, whichever is longer, prior to Screening

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2026-05-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 48 in the sum of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II score and Part III score [Efficacy] | From baseline to Week 48
  Change from Baseline to Week 48 in the sum of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II score and Part III score assessed in the practically defined OFF state. MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of four parts. Part II assesses motor experiences of daily living (Range 0-52). It contains 13 questions which are to be rated by the patient and/or caregiver. Part III assesses the motor signs of PD and is rated by the investigator (Range 0-132). Part III contains 33 scores based on 18 items. For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicates more severe symptoms of PD.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and tolerability] | From baseline to Week 48
  Incidence, nature, relationship to investigational product (IP), and severity of adverse events (AEs); Incidence of clinically significant findings for clinical laboratory evaluations, physical and neurological examinations, body weight , vital signs measurements, 12-lead o 12-lead electrocardiograms (ECGs), Columbia Suicide Severity Rating Scale (C-SSRS)
Change from Baseline to Week 48 in the MDS-UPDRS Part II score [Effect on motor function] | From baseline to Week 48
  Change from Baseline to Week 48 in the MDS-UPDRS Part II score. MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of four parts. Part II assesses motor experiences of daily living (Range 0-52). It contains 13 questions which are to be rated by the patient and/or caregiver. A higher score indicates more severe symptoms of PD.
Change from Baseline to Week 48 in the MDS-UPDRS Part III score [Effect on motor function] | From baseline to Week 48
  Change from Baseline to Week 48 in the MDS-UPDRS Part III score assessed in the practically defined OFF state. MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of four parts. Part III assesses the motor signs of PD and is rated by the investigator (Range 0-132). Part III contains 33 scores based on 18 items. For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicates more severe symptoms of PD.
Change from Baseline to Week 48 in the Timed Up and Go (TUG) test [Effect on motor function] | From baseline to Week 48
  Change from Baseline to Week 48 in the Timed Up and Go (TUG) test performed in the practically defined OFF state. The TUG is a clinical test for assessing functional mobility and balance, where a person times how long it takes to stand up from a chair, walk 3 meters, turn 180 degrees, walk back, and sit down again. A time of less than 14 to 15 seconds indicates good mobility, while longer times suggest an increased risk of falling, poor physical performance, and potentially neurological issues.
Change from Baseline to Week 48 in the Parkinson's Disease Questionnaire 39 (PDQ-39) score [Effect on quality of life] | From baseline to Week 48
  Change from Baseline to Week 48 in the Parkinson's Disease Questionnaire 39 (PDQ-39) score. The PDQ-39 is a 39-item self-report questionnaire, which assesses PD-specific health-related quality over the last month. The questionnaire measures 39 items, which assess 8 domains of health: mobility (10 items), activities of daily living (6 items), emotional well being (6 items), stigma (4 items), social support (3 items), cognitions (4 items), communication (3 items), and bodily discomfort (3 items). Each item is scored on the following scale: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, and 4 = always. Items in each subscale and the total scale can be summarized into an index and transformed linearly to a scale from 0 (perfect health as assessed by the measure) to 100 (worst health as assessed by the measure).
Change from Baseline to Week 48 in the Schwab and England Activities of Daily Living (SEADL) scale [Effect on activities of daily living] | From baseline to Week 48
  Change from Baseline to Week 48 in the Schwab and England Activities of Daily Living (SEADL) scale. The SEADL Scale assesses the capabilities of people with impaired mobility in a range of life activities. The scale uses a percentage score to rate a person's abilities, with 100% indicating complete independence (able to do all chores without slowness, difficulty, or impairment) and 0% indicating full dependence (bedridden and almost completely comatose).
Change from Baseline to Week 48 in the Patient Global Impression Scale - Severity (PGI-S) | From baseline to Week 48
  Change from Baseline to Week 48 in the Patient Global Impression Scale - Severity (PGI-S). The PGI-S is a simple, direct, easy to use scales used to rate the response of a condition to a therapy. It is a transition scale for the participant to rate their condition now as compared with how it was prior to before starting the treatment on a scale from 1 "Very much better" to 7 "Very much worse" with lower scores indicating greater improvement.
Change from Baseline to Week 48 in the Clinical Global Impressions Scale - Severity (CGI-S) | From baseline to Week 48
  Change from Baseline to Week 48 in the Clinical Global Impressions Scale - Severity (CGI-S). The CGI-C scale is a clinician-rated measures of severity of a symptom or condition, using a single item, 6-point-scale. The CGI-S scale ranges from 1 ("None") to 6 ("Very Severe") with lower scores indicating lower severity.

OTHER OUTCOMES:
Change from Baseline to Week 48 in the MDS-UPDRS Part I score [Effect on non-motor symptoms of PD] | From baseline to Week 48
  Change from Baseline to Week 48 in the MDS-UPDRS Part I score. The MDS-UPDRS is a multimodal scale consisting of four parts. Part I assesses non-motor experiences of daily living and has 2 components (Range 0-52). Part IA contains 6 questions and are assessed by the examiner (Range 0-24). Part IB contains 7 questions on non-motor experiences of daily living to be completed by the participant (Range 0-28). For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicates more severe symptoms of PD.
Change from Baseline to Week 48 in the Cognitive Summary Score (CSS) [Effect on non-motor symptoms of PD] | From baseline to Week 48
  Change from Baseline to Week 48 in the Cognitive Summary Score (CSS). The CSS is a composite score that combines results from several detailed neuropsychological tests into a single, more sensitive measure of cognitive ability. It compares the score to norms to identify deficit in cognitive areas like processing speed, working memory, and verbal memory, and tracks cognitive changes over time. CSS scores can range from 0 to 100. A lower score indicates more significant cognitive impairment.
Change from Baseline to Week 48 in the Purdue Pegboard Test (PPT) total score | From baseline to Week 48
  Change from Baseline to Week 48 in the Purdue Pegboard Test (PPT) total score performed in the practically defined OFF state. The PPT is a standardized test to assess fine and gross motor skills and coordination, commonly used to evaluate manual abilities. It measures the ability to move the arms, hands, and fingers quickly and accurately by placing pegs into a board, both with individual hands and with both hands simultaneously, and in an assembly task. The time and the number of pegs inserted is recorded. A faster time is indicative of a better function, i.e., a higher score (more pegs) signifies better performance.
Change from Baseline to Week 48 in the Geriatric Depression Scale 15-item version (GDS-15) | From baseline to Week 48
  Change from Baseline to Week 48 in the Geriatric Depression Scale 15-item version (GDS-15). The 15-item Geriatric Depression Scale (GDS-15) is a depression screening tool developed for use in older adults. The GDS-15 has a yes-no format. Scores range from 0 to 15; the higher the score the more likely the individual is experiencing depression.
Change from Baseline to Week 48 in the Movement Disorder Society-Non-motor Scale (MDS-NMS) score | From baseline to Week 48
  Change from Baseline to Week 48 in the Movement Disorder Society-Non-motor Scale (MDS-NMS) score. The MDS-NMS is a 52-item rater-administered scale to assess a wide range of non-motor symptoms in Parkinson's disease.
  It measures both frequency (0/never to 4/ >51% of the time) and severity (0/not present to 4/major distress or disturbance) of 13 domains (depression, anxiety, apathy, psychosis, impulse control/related disorders, cognition, orthostatic hypotension, urinary, sexual, gastrointestinal, sleep/wakefulness, pain, and other). Each question is scored by multiplying frequency x severity. All question scores for each domain are summed, and the scores for each domain are summed to provide the Total Score (range = 0-832) with the higher score indicating greater non-motor symptom burden. The higher the total score, the more progressed (i.e., worse) is the disease state.
Change from Baseline to Week 48 in Neuronal Synuclein Disease (NSD) stage | From baseline to Week 48
  Change from Baseline to Week 48 in Neuronal Synuclein Disease (NSD) stage. The NSD41 is a research framework that classifies the stages of diseases like PD by combining biological markers and functional impairment. It uses a 7-stage system, beginning with Stage 0 for a genetic variant and progressing through stages based on the presence of abnormal α synuclein protein, dopaminergic dysfunction, and the increasing severity of functional impairment in later stages. Higher stages are indicative of more severe functional impairment.
Number of participants who require an increase in, or initiation of, dopaminergic treatment | From baseline to Week 48
  Number of participants who require an increase in, or initiation of, dopaminergic treatment by Week 48.
Change from Baseline to Week 48 in the University of Pennsylvania Smell Identification Test (UPSIT) [Olfaction] | From baseline to Week 48
  Change from Baseline to Week 48 in in olfaction as measured with the University of Pennsylvania Smell Identification Test (UPSIT) The UPSIT is considered to be an reliable and accurate tool for diagnosing smell loss and screening for conditions like PD. The test is a 40-item, self-administered "scratch-and-sniff" test to quantitatively measure olfactory function. The test involves scratching a strip to release an odor and selecting the correct identification from multiple-choice options. The UPSIT has a minimum score of 0 and maximum score of 40 with lower scores indicating a greater degree of impairment.
Mean trough plasma levels of GT-02287 | From baseline to Week 48
  Mean concentration of GT-02287 24 hours postdose, immediately before the next dose
Mean peak plasma levels of GT-02287 | From baseline to Week 48
  Mean concentration of GT-02287 around Cmax/time to maximum concentration (Tmax)
Mean CSF levels of GT-02287 at Week 48 | Week 48
  Postdose (approximately 4 hours postdose) concentration of GT-02287 in CSF at Week 48
Changes in mechanistic and disease biomarkers | From baseline to Week 48
  Change in biomarkers in biofluids (CSF, blood, plasma) from Baseline to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Hannestad, CMO, Study Director — Gain Therapeutics, Inc.

IPD SHARING:
Plan to Share IPD: No